CLINICAL TRIAL: NCT03590847
Title: Time to Eat Study - Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB201801293
Record Dates: First submitted 2018-06-08; First posted 2018-07-18 (Actual); Results first posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Overweight
Keywords: Intermittent fasting; Inflammation; Diet; Lifestyle; Eating habits; Time Restricted Feeding
MeSH Terms: conditions — Overweight; Intermittent Fasting; Inflammation; Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intermittent fasting (Experimental): Study participants will be asked to fast for a target of 16 hours per day for a period of 4 weeks.
  Interventions: Behavioral: Intermittent Fasting

INTERVENTIONS:
Behavioral: Intermittent Fasting — Study participants will be asked to fast for a target of 16 hours per day for a period of 4 weeks. Participants will be allowed to consume calorie-free beverages, water, tea, black coffee or sugar-free gum during the fasting period. Participants will be asked to record the time of first and final food/drink consumption each day.
  Other Names: Time Restricted Feeding

SUMMARY:
The goals of this pilot study is to evaluate the safety and feasibility of time restricted feeding in an older adult population.

DETAILED DESCRIPTION:
For this 4-week pilot study, the study team will recruit 10 overweight, older adults who are at risk for, or have, mobility impairment, as measured by slow gait speed and self-reported mobility difficulty and self-reported sedentary lifestyle. All participants will receive the time restricted feeding intervention, which will consist of limiting the time in which food is consumed to 8 hours per day and fasting for 16 hours per day. The study will also assess the variance of inflammatory markers, walking speed, physical and cognitive function, grip strength, body measurements, perceived fatigability, health related quality of life and activity level. This allows the refinement of the design, recruitment yields, target population, adherence, retention, and tolerability of a larger scale study.

ELIGIBILITY:
Inclusion Criteria:

* Consent to participate in the study
* Men and women ≥ 65 years old
* Self-reported difficulty walking ¼ mile or climbing a flight of stairs
* Self-reported sedentariness (<30 minutes structured exercise per week)
* Walking speed <1 m/sec on the 4 m walk test
* Able to walk unassisted (cane allowed)
* Have a body mass index between 25 - 40 kg/m2 (inclusive)

Exclusion Criteria:

* Current dietary habits

  * Fasting >12 hours per day
  * Actively trying to lose weight by participating in formal weight loss program or significantly restricting calorie intake
  * Weight loss > 5 lbs in the past month
* Medical history or conditions

  * Resting heart rate of >120 beats per minute, systolic blood pressure > 180 mmHg or diastolic blood pressure of > 100 mmHg
  * Unstable angina, heart attack or stroke in the past 3 months
  * Continuous use of supplemental oxygen to manage a chronic pulmonary condition or heart failure
  * Rheumatoid arthritis, Parkinson's disease or currently on dialysis
  * Active treatment for cancer in the past year
  * Insulin dependent diabetes mellitus
* Taking medications that preclude fasting for 16 hours (e.g. must be taken with food at least 12 hours apart)
* Any condition that in the opinion of the investigator would impair ability to participate in the trial

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-06-28 (Actual); Primary Completion 2018-09-05 (Actual); Study Completion 2018-09-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Anton, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida Institute on Aging, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the general population in the North/Central Florida area through mailing, advertisements, and targeted outreach to individuals who have consented to participation in the Claude D. Pepper Recruitment Registry.
Pre-assignment Details: Participants were overweight, sedentary older adults (≥65 years) with mild to moderate functional limitations. Participants were excluded from the study if they were unwilling to consent or had underlying health conditions that would cause personal risk as a result of participating. A telephone screening to ensure eligibility and review protocol for obtained consent. Baseline measurements and blood samples were collected to further determine eligibility.
Period: Overall Study
Arm/Group | Intermittent Fasting
Started | 10
Completed | 9
Not Completed | 1

BASELINE CHARACTERISTICS:
Population: Overweight, sedentary older adults (≥65 years) with mild to moderate functional limitations.
Arm/Group | Intermittent Fasting
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 10
Age, Continuous [Mean (Full Range); unit: years] | 77.1 [65 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10
Body Weight [Mean (Standard Deviation); unit: kg] — Measured following the removal of excess clothing and shoes with a calibrated scale (Detecto).
  kg | 96.96 (16.2)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 34.1 (3.3)
Waist Circumference [Mean (Standard Deviation); unit: cm] — Taken at the mid-point between the participant's lowest rib and the top of his/her hip bone.
  cm | 109.43 (12.9)
Blood Glucose [Mean (Standard Deviation); unit: mg/dL] — Blood was drawn at a fasted state. Glucose levels were measured by Quest Diagnostic Clinical Laboratories, which is accredited by the College of American Pathologists.
  mg/dL | 105.6 (28.2)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] — Resting blood pressure was taken after participants spent 5 min seated in a quiet room, free of distractions. Blood pressure was obtained according to standardized protocol. Three readings of blood pressure, spaced one minute apart, were taken using a sphygmomanometer with appropriate cuff size. First reading was discarded and last two readings were averaged. If large differences were observed between second and third readings, an additional reading was taken and the median value of the three trials was used.
  mmHg | 145.9 (15.6)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] — Resting blood pressure was taken after participants spent 5 min seated in a quiet room, free of distractions. Blood pressure was obtained according to standardized protocol. Three readings of blood pressure, spaced one minute apart, were taken using a sphygmomanometer with appropriate cuff size. First reading was discarded and last two readings were averaged. If large differences were observed between second and third readings, an additional reading was taken and the median value of the three trials was used.
  mmHg | 78.1 (12.4)
Six Minute Walk Test (meters) [Mean (Standard Deviation); unit: meters] — Measures the amount of distance the participant can complete on a standard walking course in six minutes without running or overexerting themselves. Participants were instructed to walk at a fast pace and the distance covered in meters was measured.
  meters | 301.8 (91.0)
Six Minute Walk Test (m/s) [Mean (Standard Deviation); unit: m/s] — Measures the amount of distance the participant can complete on a standard walking course in six minutes without running or overexerting themselves. Participants were instructed to walk at a fast pace and the distance covered in meters was measured.
  m/s | 0.88 (0.2)
Grip Strength [Mean (Standard Deviation); unit: kg] — Participants were asked to squeeze the dynamometer as hard as possible with their dominant hand. Two measurements were taken, and the average was used in analyses. Isometric hand grip strength is a commonly used measure of upper body skeletal muscle function and is widely used as a general indicator of functional status.
  kg | 22.3 (7.0)
12-Item Short Form Survey Physical Function [Mean (Full Range); unit: units on a scale] — Summary score of the short-form physical health status from the 12-item health questionnaire, used to assess several domains of health related quality of life (HQRoL). Scores on this measure ranging from 0 to 100, with greater scores representing better health.
  units on a scale | 13.6 [9 to 18]
12-Item Short Form Survey Mental Function [Mean (Full Range); unit: score on a scale (0-100)] — Summary score of the short form mental health status from the 12-item health questionnaire, used to assess several domains of health related quality of life (HQRoL). Scores on this measure ranging from 0 to 100, with greater scores representing better health.
  score on a scale (0-100) | 22.0 [19 to 25]
12-Item Short Form Survey Total Score [Mean (Full Range); unit: score on a scale (0-100)] — Overall short form general health perception from the 12-item health questionnaire, used to assess several domains of health related quality of life (HQRoL). Scores on this measure ranging from 0 to 100, with greater scores representing better health.
  score on a scale (0-100) | 35.6 [29 to 42]
Fatigability (Mental) [Mean (Full Range); unit: score on a scale (0-50)] — The Pittsburgh Fatigability Scale is a 26-item self-administered questionnaire to measure perceived mental and physical fatigability. Scores range from 0-50 on a scale where higher scores represent higher levels of fatigability.
  score on a scale (0-50) | 13.8 [0 to 26]
Fatigability (Physical) [Mean (Full Range); unit: score on a scale (0-50)] — The Pittsburgh Fatigability Scale is a 26-item self-administered questionnaire to measure perceived mental and physical fatigability. Scores range from 0-50 on a scale where higher scores represent higher levels of fatigability.
  score on a scale (0-50) | 24.7 [11 to 32]
Cognitive Function [Mean (Full Range); unit: units on a scale] — The Montreal Cognitive Assessment (MoCA) is a 30-point tool designed to assess mild cognitive impairment. It evaluates various cognitive domains, including attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation. The total score is obtained by summing the individual subscores, with a minimum score of 0 and a maximum score of 30. Higher scores indicate better cognitive function. To minimize learning effects from repeated administrations, different versions of the test were used at baseline and week four.
  units on a scale | 25.6 [19 to 29]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events as a Measure of Safety and Tolerability
Description: At each follow-up contact (either by phone or in person), participants are asked about any changes to their health or physical function since the previous contact. The changes are documented on the adverse event log.
Time Frame: Week 4
Measure: Count of Participants; unit: Participants
Arm/Group | Intermittent Fasting
Number analyzed (Participants) | 10
Participants | 3

2. Primary Outcome: Adherence
Description: Adherence to the study intervention is measured using food intake time diary. Participants are considered compliant to the study intervention if he/she fasts between 14 - 18 hours per day for the duration of the 4 week study.
Time Frame: Week 4
Measure: Mean (Full Range); unit: percentage of days adherent
Arm/Group | Intermittent Fasting
Number analyzed (Participants) | 10
percentage of days adherent | 84 [50 to 100]

3. Primary Outcome: Retention
Description: Number of Participants who dropped out before the Week 4 clinic visit was completed.
Time Frame: Week 4
Measure: Count of Participants; unit: Participants
Arm/Group | Intermittent Fasting
Number analyzed (Participants) | 10
Participants | 1

4. Primary Outcome: Recruitment Yields
Description: Recruitment yields is measured by the number of individuals who were assessed at phone screening.
Time Frame: Baseline
Measure: Number; unit: participants
Arm/Group | Intermittent Fasting
Number analyzed (Participants) | 10
participants | 65

5. Secondary Outcome: Body Weight
Description: Body weight will be measured following the removal of excess clothing and shoes with calibrated scales. Primary study outcomes include final weight at the 4 week assessment visit.
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Intermittent Fasting
Number analyzed (Participants) | 9
kg | 94.81 (16.9)

6. Secondary Outcome: Body Mass Index (BMI)
Description: Measure of body fat using weight from previous weight measurement.
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Intermittent Fasting
Number analyzed (Participants) | 9
kg/m^2 | 33.2 (3.2)

7. Secondary Outcome: Waist Circumference
Description: Waist circumference is taken at the mid-point between the participant's lowest rib and the top of his/her hip bone.
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Intermittent Fasting
Number analyzed (Participants) | 9
cm | 109.23 (12.3)

8. Secondary Outcome: Blood Glucose
Description: Blood was drawn at a fasted state. Glucose levels were measured by Quest Diagnostic Clinical Laboratories, which is accredited by the College of American Pathologists.
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Intermittent Fasting
Number analyzed (Participants) | 9
mg/dL | 107.3 (29.4)

9. Secondary Outcome: Systolic Blood Pressure
Description: Resting blood pressure was taken after participants spent 5 min seated in a quiet room, free of distractions. Blood pressure was obtained according to standardized protocol. Three readings of blood pressure, spaced one minute apart, were taken using a sphygmomanometer with appropriate cuff size. First reading was discarded and last two readings were averaged. If large differences were observed between second and third readings, an additional reading was taken and the median value of the three trials was used.
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Intermittent Fasting
Number analyzed (Participants) | 9
mmHg | 148.22 (24.2)

10. Secondary Outcome: Diastolic Blood Pressure
Description: as for outcome 9
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Intermittent Fasting
Number analyzed (Participants) | 9
mmHg | 78.89 (8.3)

11. Secondary Outcome: 6 Minute Walk Test (Meters)
Description: The 6-Minute Walk Test (6MWT) measures the distance a participant can walk on a standard course within six minutes, without running or overexerting themselves. Contraindications for test administration and stopping rules will be followed according to the guidelines of the American Thoracic Society. The outcome will be reported in meters (m), representing the total distance covered during the 6-minute walk.
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Intermittent Fasting
Number analyzed (Participants) | 9
meters | 310.89 (111.2)

12. Secondary Outcome: 6 Minute Walk Test (m/s)
Description: The 6 Minute Walk test measures the amount of distance the participant can complete on a standard walking course in six minutes without running or overexerting themselves. Contraindications for test administration and stopping rules based on American Thoracic Society will be followed. Walking speed was calculated by dividing number of meters walked by total time completed (360 seconds/6 minutes).
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Intermittent Fasting
Number analyzed (Participants) | 9
m/s | 0.92 (0.2)

13. Secondary Outcome: Grip Strength (Dominant Hand)
Description: Isometric hand grip strength is a commonly used measure of upper body skeletal muscle function and has been widely used as a general indicator of functional status.Total force output is reported in kilograms (kg).
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Intermittent Fasting
Number analyzed (Participants) | 9
kg | 24.0 (6.8)

14. Secondary Outcome: 12-Item Short Form Survey Physical Function (Summary Score)
Description: Self-administered, 12-item questionnaire to measure health-related quality of life. Short form (SF) physical health status with scores on this measure ranging from 0 to 100, where greater scores represent better health.
Time Frame: Week 4
Measure: Mean (Full Range); unit: score on a scale (0-100)
Arm/Group | Intermittent Fasting
Number analyzed (Participants) | 9
score on a scale (0-100) | 14.9 [12 to 18]

15. Secondary Outcome: 12-Item Short Form Survey Mental Function (Summary Score)
Description: Self-administered, 12-item questionnaire to measure health-related quality of life. Short form (SF) mental health status with scores on this measure ranging from 0 to 100, where greater scores represent better health.
Time Frame: Week 4
Measure: Mean (Full Range); unit: score on a scale (0-100)
Arm/Group | Intermittent Fasting
Number analyzed (Participants) | 9
score on a scale (0-100) | 22.8 [20 to 25]

16. Secondary Outcome: 12-Item Short Form Survey Total Score
Description: A self-administered, 12-item questionnaire is used to measure health-related quality of life, specifically the Short Form (SF) general health perception. Scores range from 0 to 100, with higher scores indicating better perceived health. Total scores are reported.
Time Frame: Week 4
Measure: Mean (Full Range); unit: score on a scale (0-100)
Arm/Group | Intermittent Fasting
Number analyzed (Participants) | 9
score on a scale (0-100) | 37.7 [34 to 42]

17. Secondary Outcome: Fatigability Questionnaire (Mental Subscale)
Description: A self-administered, 26-item questionnaire to measure perceived mental and physical fatigability. Scores range from 0-50 on a scale where higher scores represent higher levels of fatigability.
Time Frame: Week 4
Measure: Mean (Full Range); unit: score on a scale (0-50)
Arm/Group | Intermittent Fasting
Number analyzed (Participants) | 9
score on a scale (0-50) | 14.7 [0 to 28]

18. Secondary Outcome: Fatigability Questionnaire (Physical Subscale)
Description: as for outcome 17
Time Frame: Week 4
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Intermittent Fasting
Number analyzed (Participants) | 9
score on a scale | 24.9 [10 to 35]

19. Secondary Outcome: Montreal Cognitive Assessment
Description: The Montreal Cognitive Assessment (MoCA) is a 30-point tool designed to assess mild cognitive impairment. It evaluates various cognitive domains, including attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation. The total score is obtained by summing the individual subscores, with a minimum score of 0 and a maximum score of 30. Higher scores indicate better cognitive function. To minimize learning effects from repeated administrations, different versions of the test were used at baseline and week four.
Time Frame: Week 4
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Intermittent Fasting
Number analyzed (Participants) | 9
score on a scale | 25.9 [20 to 29]

20. Secondary Outcome: Circulating (Plasma) microRNA
Description: The fold change in circulatory microRNA post-TRE regimen will be measured using the HTG EdgeSeq miRNA Whole Transcriptome Assay, which profiles the expression of circulatory miRNAs. The total number of differentially expressed miRNAs will be analyzed, including a breakdown of how many were differentially upregulated and downregulated.
Time Frame: Week 4
Measure: Number; unit: Number of Differentially Expressed miRNA
Arm/Group | Intermittent Fasting
Number analyzed (Participants) | 9
Number of Differentially Expressed miRNA
  Differentially expressed miRNA (total) | 14
  Differentially expressed miRNA (downregulated) | 8
  Differentially expressed miRNA (upregulated) | 6

ADVERSE EVENTS:
Time Frame: Baseline to Week 4
Arm/Group | Intermittent Fasting
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 3/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intermittent Fasting (N=10)
Headache (Nervous system disorders) | 2 — Participants reported headaches during fasting periods.
Dizziness (Ear and labyrinth disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-07-06): https://cdn.clinicaltrials.gov/large-docs/47/NCT03590847/Prot_SAP_000.pdf
  • Informed Consent Form (2018-06-27): https://cdn.clinicaltrials.gov/large-docs/47/NCT03590847/ICF_001.pdf